CLINICAL TRIAL: NCT00002361
Title: A Multicenter, Open-Label, 24-Week Study to Evaluate the Safety and Activity of Indinavir Sulfate 800 Mg b.i.d. in Combination With Ritonavir 200 Mg b.i.d. and Two NRTIs in HIV-1 Infected Patients Who Failed PI Therapy
Brief Title: Safety and Effectiveness of an Anti-HIV Drug Combination in HIV-Positive Patients Who Have Failed Previous Treatment With Protease Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 246S; 088-00
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Indinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir

SUMMARY:
The purpose of this study is to see if it is safe and effective to give an anti-HIV drug combination containing indinavir and ritonavir to HIV-positive patients who have failed previous treatment with protease inhibitors.

DETAILED DESCRIPTION:
Patients receive indinavir and ritonavir twice daily plus 2 NRTIs (NRTIs are not provided by this study). Physical examinations and laboratory tests, including plasma viral RNA levels and CD4 cell counts, are performed at Day 1 and Weeks 4, 8, 12, 16, 20, and 24 (or at discontinuation). The incidence of serious and drug-related adverse experiences is tabulated to determine drug safety. The proportion of patients achieving plasma viral RNA levels below 50 copies/ml (by UltraSensitive assay) are estimated statistically to determine drug efficacy.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a viral load (level of HIV in the blood) of 2500 copies/ml or greater within 45 days of study entry.
* Have a CD4 cell count of 100 cells/mm3 or greater within 45 days of study entry.
* Have been on an anti-HIV drug regimen containing a protease inhibitor for at least 16 weeks and initially did well on this treatment (your viral load decreased significantly) but later experienced treatment failure on this drug combination (your viral load increased significantly).
* Experienced treatment failure within 24 weeks of study entry.
* Are 18 years of age or older.
* Agree to use effective barrier methods of birth control (such as condoms) during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Are allergic to ritonavir or indinavir.
* Have hepatitis.
* Have an abnormal chest x-ray or abnormal liver function tests.
* Have taken 2 protease inhibitors at the same time for 7 or more days.
* Have taken non-nucleoside reverse transcriptase inhibitors (NNRTIs) in the 2 weeks before study entry.
* Have a medical condition that might make it unsafe for you to take the study drugs.
* Have experienced resistance to NRTIs and no new NRTI therapy is possible.
* Have taken certain medications.
* Abuse alcohol or drugs.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - LAC / USC Med Ctr / Infectious Diseases, Los Angeles, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ / Div of Infect Diseases, Chicago, Illinois
  - Chase Braxton Health Service, Baltimore, Maryland
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Albany Med College, Albany, New York
  - Univ of North Carolina / Infectious Disease Division, Chapel Hill, North Carolina
  - The Research and Education Group, Portland, Oregon